CLINICAL TRIAL: NCT00001722
Title: Adipose Tissue Microperfusion to Assess Leptin Secretion and Its Relations With Lipolysis in Humans
Brief Title: Fat Tissue Microperfusion to Measure Leptin Secretion and Its Relations With Fat Breakdown in Humans
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980103; 98-CH-0103
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-07

CONDITIONS: Healthy; Obesity
Keywords: Obesity; Sympathetic Nervous System; Fat Tissue; Metabolism; Adipose Tissue; Microdialysis; Leptin; Lipolysis; Normal Volunteer
MeSH Terms: conditions — Obesity

SUMMARY:
Leptin is a hormone that acts in the body as a chemical messenger. It is produced in fat cells and is believed to regulate body weight in humans. Leptin decreases appetite and influences the energy balance of the body.

This study will attempt to measure levels of leptin production in the fat pad of the body by using a process called microperfusion. Microperfusion works by inserting 2 to 3 probes (thin tubes) into the fat pad around the belly button. These probes can measure chemicals in an area known as the extracellular space. This is the small space between cells and blood vessels that hormones, medicines, nutrients, and salts travel through.

The study will investigate the effects of a meal, insulin, glucose (sugar), and the medication isoproterenol on leptin levels. Researchers believe that leptin levels are regulated along with the enzyme, hormone sensitive lipase (HSL). When hormone sensitive lipase is activated fat is broken down in a process called lipolysis. In addition, increased levels of HSL result in decreased levels of leptin, which in turn increases appetite and food intake.

DETAILED DESCRIPTION:
The adipocyte hormone leptin serves as a humoral signal of energy stores, acting on central neuronal networks that regulate ingestive behavior and energy balance. The basis for the circadian rhythm and pulsatility of circulating leptin levels in the face of a relatively stable adipose mass is not known. We have already established the feasibility and validity of adipose tissue microperfusion in humans for measurements of leptin in adipose tissue interstitial fluid. The aim of this study now is to assess the specific aspects of the regulation of adipose tissue metabolism in situ.

The hormone sensitive lipase (HSL) catalyzes the final, rate limiting step of energy mobilization from adipose tissue. Its activation results in hydrolysis of triglycerides, a process referred to as lipolysis. Increased HSL activity during fasting and stress, is physiologically coupled with significant reductions in circulating leptin levels, which in turn, results in increased food intake, and thus, restoration of energy balance. We hypothesize that local neural signals from the sympathetic nervous system to adipocytes through beta-adrenergic receptors simultaneously regulate leptin secretion and lipolysis, the latter via the modulation of HSL activity. This hypothesis will be tested by measurements of interstitial levels of leptin and glycerol in adipose tissue in situ before and after local administration of a beta-adrenergic agonist. Food intake and beta-adrenergic stimulation are excellent potential stimuli in the study of the novel fat-derived hormones, resistin and adiponectin.

We hypothesize that insulin has regulatory effects on leptin secretion and lipolysis. This hypothesis will be tested by measurement of interstitial levels of leptin, TNF-alpha, and interleukin-6 in adipose tissue in situ and after local administration of insulin.

ELIGIBILITY:
INCLUSION CRITERIA

Healthy subjects ages 18 to 50 years.

Healthy volunteers studied as outpatients.

EXCLUSION CRITERIA

Minors (less than 18 years of age)

Subjects taking any medication on a regular basis.

Individuals with hepatic, renal, HPA axis or thyroid dysfunction.

Very lean individuals (defined as a body mass index less than 19).

Smokers.

Pregnant or lactating woman.

Individuals with allergies to teflon, polyethylene or skin tape.

Individuals with known allergy to isoproterenol.

Individuals unable to abstain from alcohol, tobacco, tea, and coffee for 18 hours prior and during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 1998-04; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Zhang Y, Proenca R, Maffei M, Barone M, Leopold L, Friedman JM. Positional cloning of the mouse obese gene and its human homologue. Nature. 1994 Dec 1;372(6505):425-32. doi: 10.1038/372425a0. PMID 7984236
- [Background] Campfield LA, Smith FJ, Burn P. The OB protein (leptin) pathway--a link between adipose tissue mass and central neural networks. Horm Metab Res. 1996 Dec;28(12):619-32. doi: 10.1055/s-2007-979867. PMID 9013731
- [Background] Caro JF, Sinha MK, Kolaczynski JW, Zhang PL, Considine RV. Leptin: the tale of an obesity gene. Diabetes. 1996 Nov;45(11):1455-62. doi: 10.2337/diab.45.11.1455. No abstract available. PMID 8866547